CLINICAL TRIAL: NCT04432038
Title: Healthy Lifestyle or Pro-health Obsession During the Pandemic - a Multinational Study
Brief Title: Healthy Lifestyle or Pro-health Obsession During the Pandemic
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Gdansk University of Physical Education and Sport (Other)
Collaborators: University Hospital of Split (Other); University of Gondar (Other); Universidad Pablo de Olavide (Other); Universitas Padjadjaran (Other); University of Social Welfare and Rehabilitation Science (Other); DPFA Academy of Work and Health, Leipzig (Unknown); Instituto Piaget (Other); University of Peradeniya (Other); Catholic University of the Sacred Heart (Other); University of Évora (Other); Norwegian School of Sport Sciences (Other); Klaipėda University (Other); Universitatea Alexandru Ioan Cuza (Unknown); Institut Catholique de Paris (Unknown); University of Gdansk (Other); Jagiellonian University (Other); International University of Business Agriculture and Technology (Unknown); Beijing Sport University (Other); University of Nigeria, Enugu Campus (Other); University of Sargodha (Other); University of Brasilia (Other); Wright State University (Other); Vietnam National University (Other); Taras Shevchenko National University of Kyiv (Other); Astana Medical University (Other); International Islamic Academy of Uzbekistan (Unknown); Menoufia University (Other); Zhengzhou University (Other)
Responsible Party: Sponsor
Other Study IDs: GdanskUPES
Record Dates: First submitted 2020-06-07; First posted 2020-06-16 (Actual); Last update posted 2021-04-09 (Actual); Status verified 2020-06

CONDITIONS: Adult; Global Health
Keywords: COVID-19; well-being; physical activity; nutrition; body image
MeSH Terms: conditions — COVID-19; Motor Activity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (28):
- General population of adults from about 30 countries: Data will be collected in general population of adults from about 30 countries. Questionnaires contain also questions about the occurrence of chronic illnesses, being a professional athlete, etc. to control all such aspects.
- General population of adults from Poland
- General population of adults from Germany
- General population of adults from China
- General population of adults from Vietnam
- General population of adults from Spain
- General population of adults from Brazil
- General population of adults from Croatia
- General population of adults from Ethiopia
- General population of adults from France
- General population of adults from Indonesia
- General population of adults from Iran
- General population of adults from Sri Lanka
- General population of adults from USA
- General population of adults from Italy
- General population of adults from South Africa
- General population of adults from Portugal
- General population of adults from Norway
- General population of adults from Lithuania
- General population of adults from Romania
- General population of adults from Pakistan
- General population of adults from Ukraine
- General population of adults from India
- General population of adults from Japan
- General population of adults from Russia
- General population of adults from Bangladesh
- General population of adults from Nigeria
- General population of adults from Egypt

SUMMARY:
Citizens of many countries are in the high peak period of the outbreak of the COVID-19 virus. People are currently struggling with the total cessation of certain aspects of normal life. The situation associated with the pandemic can lead to the development of many problems connected both with mental and physical health. The investigators, as psychologists, would like to better understand this difficult situation and identify mechanisms which can lead to health problems. Therefore, group of researchers and practitioners created this study to investigate how people in general cope with this critical situation. The researchers would like to estimate the following variables which participants will evaluate before and during the pandemic period: levels of physical activity, attitudes towards one's body, attitudes towards eating, and psychological well-being. The investigators would like to involve experts and scientists from all around the world. Through this research and by investigating how people cope with this critical situation the solutions for psychological care and interventions for global crisis situations like the COVID-19 pandemic might be identified.

ELIGIBILITY:
Inclusion Criteria:

- Age: min 18 years old

Exclusion Criteria:

- no

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: The investigators will approach individuals from Bangladesh, Brazil, China, Croatia, Ethiopia, France, Germany, Indonesia, Iran, Italy, Lithuania, Nigeria, Norway, Pakistan, Portugal, Romania, South Africa, Spain, Sri Lanka, USA, Vietnam
Sampling Method: Non-Probability Sample
Enrollment: 50000 (Estimated)
Dates: Start 2020-06-19 (Actual); Primary Completion 2021-06-19 (Estimated); Study Completion 2021-06-30 (Estimated)

PRIMARY OUTCOMES:
Levels of Physical Activity | Baseline
  measured by Inventory of Physical Activity Objectives (IPAO) by Lipowski & Zaleski is used to examine the motivating function of objectives determining one to undertake physical activity. The respondent answers questions regarding his/her involvement in competitive sports (both present and previous), and forms and intensity of his/her physical activity. The survey allows analyzing objectives in terms of their dimensions (importance, expectations, conflict), as well as dimensions of action (exercise, endurance, satisfaction). The respondent is given a (multiple) choice of objectives behind his/her physical activity. Four scales of goal-oriented behaviours associated with PA are distinguished in the test: motivational value, time management, persistence in action, motivational conflict. The higher the results of these scales - the higher the motivation to physical activity. IPAO is characterized by good psychometric properties, the Cronbach's α for IPAO reached 0,78.
Eating Attitudes | Baseline
  measured by Eating Attitudes Test (EAT-26) by Garner, Olmsted, Bohr & Garfinkel (1982). It's a self-report measure of symptoms and concerns characteristic of eating disorders. The EAT-26 can be used in a non-clinical as well as a clinical setting not specifically focused on eating disorders. Questionnaire is rated on a six-point scale based on how often the individual engages in specific behaviors. Scores greater than 20 indicate a need for further investigation by a qualified professional. Research using different EAT-26 language versions has a satisfactory Crombach's alpha 0,78-0,92.

SECONDARY OUTCOMES:
Psychological wellbeing | Baseline
  measured by Psychological Well-Being Scales (PWBS) by Ryff (2004). The PWB scales incorporate six dimensions: autonomy, positive relations with others, environmental mastery, personal growth, purpose in life and self-acceptance. Respondents rate how strongly they agree or disagree with 18 statements using a 7-point scale, higher scores indicate greater wellbeing.
Physical wellbeing | Baseline
  measured by SF-12v2 Health Survey, the SF-12v2 is a practical, reliable and valid measure of physical and mental health, it uses just 12 questions. Higher scores indicate a higher level of physical wellbeing
Obligatory Exercise | Baseline
  measured by Obligatory Exercise Questionnaire (OEQ) by Pasman & Thompson (1988). OEQ allows to measure excessive exercise activity, especially as it relates to eating disorders. The OEQ contains three factors: Emotional Element of Exercise; Exercise Frequency and Intensity; and Exercise Preoccupation. All items indicate higher endorsement of and engaging in obligatory exercise behaviors.
Attitudes Towards Body | Baseline
  measured by Sociocultural Attitudes Towards Appearance (SATAQ 3) by Thompson et al (2014) - widely used measure of societal influences on body image and eating disturbances. SATAQ 3 has subscales that assess internalization (general, athlete), pressures, and information. Items are rated on a five point response scale, with higher scores indicating greater media endorsement.
Body Image Disturbance | Baseline
  measured by Fear of Negative Appearance Evaluation Scale (FNAES) developed by Lundgren, Anderson &Thompson (2004) - an eight-item self-report measure that assesses apprehension about appearance evaluation. The higher the FNEAS score the more fear of negative appearance evaluation by others is experienced.

CONTACTS AND LOCATIONS:
Locations (1):
- Gdansk University of Physical Education and Sport, Gdansk, Poland

REFERENCES:
- [Background] Garner DM, Olmsted MP, Bohr Y, Garfinkel PE. The eating attitudes test: psychometric features and clinical correlates. Psychol Med. 1982 Nov;12(4):871-8. doi: 10.1017/s0033291700049163. PMID 6961471
- [Background] Thompson JK, van den Berg P, Roehrig M, Guarda AS, Heinberg LJ. The sociocultural attitudes towards appearance scale-3 (SATAQ-3): development and validation. Int J Eat Disord. 2004 Apr;35(3):293-304. doi: 10.1002/eat.10257. PMID 15048945
- [Background] Lundgren JD, Anderson DA, Thompson JK. Fear of negative appearance evaluation: development and evaluation of a new construct for risk factor work in the field of eating disorders. Eat Behav. 2004 Jan;5(1):75-84. doi: 10.1016/S1471-0153(03)00055-2. PMID 15000956
- [Background] Ryff CD. Psychological well-being revisited: advances in the science and practice of eudaimonia. Psychother Psychosom. 2014;83(1):10-28. doi: 10.1159/000353263. Epub 2013 Nov 19. PMID 24281296
- [Derived] Li K, Walczak-Kozlowska T, Lipowski M, Li J, Krokosz D, Su Y, Yu H, Fan H. The effect of the Baduanjin exercise on COVID-19-related anxiety, psychological well-being and lower back pain of college students during the pandemic. BMC Sports Sci Med Rehabil. 2022 Jun 8;14(1):102. doi: 10.1186/s13102-022-00493-3. PMID 35676708
- See also: Lipowski, M., Zaleski, Z. (2015). Inventory of Physical Activity Objectives (IPAO) - a new method in measuring motives for physical activity and sport. Health Psychology Report, 3(1), 47-58 — https://doi.org/10.5114/hpr.2015.49462